CLINICAL TRIAL: NCT02746601
Title: My Health eSnapshot - A Preconception Health Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellington-Dufferin-Guelph Public Health (Other Government)
Collaborators: University of Guelph (Other); Boston Medical Center (Other); East Wellington Family Health Team (Unknown); Minto-Mapleton Family Health Team (Unknown); Upper Grand Family Health Team (Unknown); Norfolk Family Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-1
Record Dates: First submitted 2016-04-10; First posted 2016-04-21 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Preconception Care; Health Information Technology; Primary Health Care; Risk Assessment
MeSH Terms: interventions — Risk Assessment; Counseling; Health Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risk Assessment, Counselling & Resources (Experimental): Patients complete an electronic preconception health risk assessment tool. Results from the tool are directly uploaded or scanned into the patients' electronic medical record. A healthcare provider provides behavioural counselling, based on results of the risk assessment. Patients are given a customized handout that includes health recommendations and resources based on the patient's identified risk factors.
  Interventions: Behavioral: Risk Assessment, Counselling & Resources

INTERVENTIONS:
Behavioral: Risk Assessment, Counselling & Resources — A risk assessment tool is completed on a tablet. The results are scanned into the patient's electronic medical record. A healthcare provider gives behavioural counselling on identified risk factors. The patient is given a customized handout that includes health recommendations and resources based on the participant's identified risk factors.

SUMMARY:
The purpose of the research is to identify the prevalence of preconception health (PCH) risk factors in the Wellington-Dufferin-Guelph (WDG) catchment area and to determine whether or not a client-driven electronic preconception health risk assessment tool "My Health eSnapshot", for use during healthcare visits, will increase preconception health knowledge and behaviour change among women of reproductive age (15-49 years).

DETAILED DESCRIPTION:
The purpose of the project is:

1. To develop a client-driven electronic preconception health client risk assessment tool for use in a primary care setting.
2. To develop a customized key message handout for patients based on their risk assessment results.
3. To determine a successful and sustainable process for healthcare providers (HCPs) to administer the risk assessment tool and discuss results with patients within their primary care setting.
4. To increase participants' knowledge of preconception health and their risk factors as a results of the risk assessment tool and discussion with their HCP.
5. To modify participants' health behaviours as a result of the risk assessment tool and discussion with their HCP.
6. To increase WDG Public Health's understanding of the most prevalent preconception health risk factors among reproductive women in WDG.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (15-49 years)
* Not pregnant and have not had a hysterectomy
* A resident of the Wellington-Dufferin-Guelph catchment area
* Able to read and write in English
* Have a valid email address
* Willing to create a unique identifier code during the study to protect their identify
* Are comfortable using a tablet

Exclusion Criteria:

-

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient-reported risk factors as assessed by Risk Assessment Tool | Baseline
  Patient completes a risk assessment tool in their healthcare provider's office on a tablet, prior to an appointment with their Health Care Provider
Patient-reported feedback on Risk Assessment, Counselling, and Resources as assessed by a One-Week Survey | One week
  The patient will complete an online survey tool in their home one week after completing the risk assessment tool. The survey asks questions about their experience competing the risk assessment tool, talking with their health care provider, and receiving their customized patient handout. The patient will also provide feedback on the strengths and limitations of the risk assessment tool and patient handout. This feedback will contribute to future modifications to study tools and processes.
Patient-reported health behaviour change and motivation for health behaviour change as assessed by a two-month survey | Two months
  Patient complete an online survey tool in their home two months after completing the risk assessment tool. The survey asks questions about whether there has been any changes in motivation regarding changing health behaviours and whether any changes have actually been made to the health behaviours.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Minto-Mapleton Family Health Team, Drayton, Ontario
  - East Wellington Family Health Team, Erin, Ontario
  - Upper Grand Family Health Team, Fergus, Ontario
  - Norfolk Family Medical, Guelph, Ontario
  - University of Guelph, Guelph, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Non-identifying, client level data will be shared with Boston Medical Centre via encrypted means.